CLINICAL TRIAL: NCT06495775
Title: Stool Sampling in the Acute Isolated Patient, Efficient Acquiring With a Novel Device
Brief Title: Stool Sampling in the Acute Isolated Patient , Efficient Acquiring With a Novel Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SJ-866
Record Dates: First submitted 2021-05-05; First posted 2024-07-11 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2024-06

CONDITIONS: Feasibility Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- admitted patients (Experimental): fecal sampling
  Interventions: Device: quickfact

INTERVENTIONS:
Device: quickfact — fecal sampling

SUMMARY:
stool sample device tested on patients admitted to oncological dept. with diarrhea, in order to shorten time in isolation and time to relevant treatment.

DETAILED DESCRIPTION:
the stool sample device will be tested on all patients admitted to an oncological dept. on Zealand University Hospital, with diarrhea, in order to examine if the the device is feasabel and able to shorten time in isolation and time to relevant treatment.

ELIGIBILITY:
Inclusion Criteria:

* Understanding Danish
* admitted to dept og oncology with diarrhea
* cognitive intact
* Co operable to fecal sampling

Exclusion Criteria:

* expected survival less than 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2025-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Dorte b Krapper, Principal Investigator — Oncological department, Zealand University Hospital
Locations (1):
- Zealand University Hospital, Roskilde, Region Sjælland, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: all 50 participants was recruited succes fully and in rolled in the study
Groups:
- Admitted Patients: fecal sampling, instant attempt of acquiring of stool sample from acute admitted patients with diarrhea with the novel device, the stool sample is collected bedside, and if an stool sample is acquired it is there after analysed with standard analysis for infectious pathogenes.
Period: Overall Study
Arm/Group | Admitted Patients
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Admitted Patients
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Denmark | 50
Number of Participants With Stool Sample Acquired and Analyzed [Number; unit: Number of Participants With Stool Sample] — sufficient amount of stool aqquired for a stool sample to be analysed
  Number of Participants With Stool Sample | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Stool Sample Acquired
Description: instant acquiring of stool sample from acute admitted patients with diarrhea, the stool sample is collected bedside, and there after analysed with standard analysis for infectious pathogenes.
Time Frame: the sample is intended to be collected in an expected time range is within 1-2 hours after admission
Measure: Count of Participants; unit: Participants
Groups:
- Admitted Patients: fecal sampling, instant acquiring of stool sample from acute admitted patients with diarrhea, the stool sample is collected bedside, and there after analysed with standard analysis for infectious pathogenes.
Arm/Group | Admitted Patients
Number analyzed (Participants) | 50
Participants | 46

2. Primary Outcome: Safety of Device
Description: sampling with out harm to patient
Time Frame: 5 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Admitted Patients
Number analyzed (Participants) | 50
Participants | 50

ADVERSE EVENTS:
Time Frame: from enrollment til end of follow up, up to 2 weeks
Arm/Group | Admitted Patients
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

LIMITATIONS AND CAVEATS:
none relevant

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT06495775/Prot_000.pdf